CLINICAL TRIAL: NCT03798678
Title: Phase I Dose-Escalation and Dose-Expansion Trial of a Novel Glutaminase Inhibitor (CB-839 HCl) in Combination With Carfilzomib and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Brief Title: CB-839 HCl in Combination With Carfilzomib and Dexamethasone in Treating Patients With Recurrent or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00111; NCI-2019-00111 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10219 (Other: Mayo Clinic Cancer Center LAO); 10219 (Other: CTEP); UM1CA186686 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CB-839 HCI, dexamethasone, carfilzomib) (Experimental): Patients receive glutaminase inhibitor CB-839 Patients receive glutaminase inhibitor CB-839 hydrochloride PO every 12 hours on days 1-28, dexamethasone PO on days 1, 2, 8, 9, 15, 16, and 23, and carfilzomib IV over 10 minutes on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Telaglenastat Hydrochloride

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Carfilnat; CFZ; Kyprolis; PR 171; PR-171; PR171
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Telaglenastat Hydrochloride — Given PO
  Other Names: CB-839 HCl; Glutaminase Inhibitor CB-839 Hydrochloride

SUMMARY:
This phase I trial studies the best dose of CB-839 HCl when given together with carfilzomib and dexamethasone in treating patients with multiple myeloma that has come back or does not respond to previous treatment. CB-839 HCl and carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CB-839 HCl, carfilzomib, and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of glutaminase inhibitor CB-839 hydrochloride (CB-839 HCl) in combination with carfilzomib and dexamethasone.

SECONDARY OBJECTIVES:

I. Evaluate the safety and tolerability of CB-839 HCl in combination with carfilzomib and dexamethasone.

II. To determine the overall response rate (ORR) associated with the combination of CB-839 HCl with carfilzomib and dexamethasone.

CORRELATIVE RESEARCH OBJECTIVES:

I. Evaluate plasma pharmacokinetic (PK) profiles of CB-839 HCl and carfilzomib when used in combination.

II. To perform molecular profiling assays on malignant and normal tissues, including, but not limited to, whole exome sequencing (WES), messenger ribonucleic acid (RNA) sequencing (RNAseq), circulating cell free (cf) deoxyribonucleic acid (DNA) analysis, flow cytometry assessments, immunohistochemical (IHC) staining, and metabolomics-based assessments in order to identify potential predictive and prognostic biomarkers, and identify resistance mechanisms using genomic DNA, RNA, flow cytometry, IHC, and metabolomics-based assessment platforms.

III. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research.

IV. To bank CD138+ multiple myeloma (MM) cells from the bone marrow, and blood (for cfDNA analysis) obtained from patients at the Experimental Therapeutics Clinical Trials Network (ETCTN) Biorepository at Nationwide Children's Hospital.

OUTLINE: This is a dose escalation study of glutaminase inhibitor CB-839 hydrochloride.

Patients receive glutaminase inhibitor CB-839 hydrochloride orally (PO) every 12 hours on days 1-28, dexamethasone PO on days 1, 2, 8, 9, 15, 16, and 23, and carfilzomib intravenously (IV) over 10 minutes on days 1, 2, 8, 9, 15, and 16. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then periodically for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed and/or refractory myeloma and be experiencing disease relapse
* Patients must have measurable disease by International Myeloma Working Group (IMWG) criteria (any of the following):

  * Serum M-protein >= 0.5 g/dL or for IgA myeloma, an elevated IgA level by quantitative IgA nephelometry
  * Urine M-protein >= 200 mg in a 24-hour collection
  * Serum free light chain level >= 10 mg/dL with an abnormal free light chain ratio
  * Measurable plasmacytoma by cross sectional imaging (computed tomography [CT], magnetic resonance imaging [MRI] or [18F]-fluorodeoxyglucose positron emission tomography with CT [FDG PET/CT])
  * 20% or more light chain restricted, clonal plasma cells in the bone marrow
* At least two prior lines of therapy and all patients should have at least been exposed to a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-CD38 antibody
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000 cells/mm3 without growth factors (within 14 days of enrollment)
* Hemoglobin >= 8 g/dL (within 14 days of enrollment)
* Platelets >= 50,000 cells/mm3 (>= 30,000 cells/mm3 if bone marrow plasma cells >= 50% at enrollment)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< institutional ULN OR glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Willingness to undergo interim bone marrow biopsy/aspiration for clinical purposes
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

  * The effects of CB-839 HCl on the developing human fetus are unknown. For this reason and because carfilzomib caused embryo-fetal toxicity in pregnant rabbits at doses lower than the recommended dose, women of child-bearing potential and men must agree to use two effective methods of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of CB-839 HCl, carfilzomib, and dexamethasone administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CB-839 HCl, carfilzomib, and dexamethasone administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are refractory or intolerant to carfilzomib (prior carfilzomib exposure accepted)
* Patients who have received recent prior chemotherapy with:

  * Alkylators (e.g., melphalan, cyclophosphamide) and anthracyclines =< 14 days prior to registration,
  * High dose corticosteroids and immunomodulatory drugs (thalidomide or lenalidomide) =< 7 days prior to registration, or
  * Monoclonal antibodies =< 14 days prior to registration
* Patients who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1 except peripheral neuropathy)
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CB-839 HCl, carfilzomib, or dexamethasone
* Patients with uncontrolled intercurrent illness
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use two effective methods of contraception from the time of signing the informed consent form through 4 months after the last dose of study drug
  * Nursing women
  * And men who are unwilling to use birth control while taking the drug and for 4 months after stopping treatment

    * Pregnant women are excluded from this study because carfilzomib is a PI with the potential for abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with CB-839 HCl, carfilzomib, and dexamethasone, breastfeeding should be discontinued if the mother is treated with this drug combination
* Adverse cardiac history (unstable angina, myocardial infarction less than 4 months, New York Heart Association [NYHA] class III or IV congestive heart failure [CHF], ejection fraction [EF] < 40%, uncontrolled arrhythmias)
* Concomitant high dose corticosteroids other than what is part of treatment protocol (concurrent use of corticosteroids). EXCEPTION: Patients may be on chronic steroids (maximum dose 10 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, e.g., adrenal insufficiency, rheumatoid arthritis, etc
* Central nervous system (CNS) involvement

  * Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs
* Concurrent amyloid light-chain (AL) amyloidosis
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has >= grade 3 peripheral neuropathy or grade 2 with pain on clinical examination during the screening period
* Major surgery within 14 days before study registration
* On concurrent treatment with an HIV protease inhibitor

  * Human immunodeficiency virus (HIV) protease inhibitors can affect the unfolded protein response in myeloma cells as well as the activity of PIs
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of CB-839 HCl including difficulty swallowing, refractory vomiting, gastric resection or bypass, or duodenal/jejunal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase II dose (RP2D) | Up to 28 days
  MTD will be determined by dose limiting toxicity (DLT). MTD is defined as the dose level below the lowest dose that induces DLT in at least 2 patients (out of 6). The highest dose is defined as the RP2D. A standard cohort 3+3 design will be used.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after study treatment
  Incidence of adverse events will be graded according to Common Terminology Criteria for Adverse Events version 5.0. The number and severity of all AEs (overall and by dose-level) will be tabulated and summarized in this patient population. These data will be summarized with and without regard to the relationship to the treatment (i.e., ignoring the relationship data and after sub-setting the data to only events that are at least possibly related to study drug).
Overall response rate (ORR) | Up to 1 year
  The ORR will be defined as the percentage of patients that achieve at least a partial response (as their best response). Properties of the binomial distribution will be used in order to construct an exact 95% confidence interval around this proportion.

OTHER OUTCOMES:
Pharmacokinetic (PK) profiles and pharmacodynamic effect | Days 1 and 15 of cycle 1
  PK and pharmacodynamic data will be examined in an exploratory manner.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson I Gonsalves, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio